CLINICAL TRIAL: NCT03023722
Title: An Open-label, Phase II Study of Intravenous Anetumab Ravtansine (BAY 94-9343), an Anti-mesothelin Antibody Drug Conjugate, in Pretreated Mesothelin-expressing Advanced Pancreatic Cancer
Brief Title: Phase II Anetumab Ravtansine in Pre-treated Mesothelin-expressing Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1608018265
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — anetumab ravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): Patients with advanced metastatic pancreatic cancer who have measurable disease
  Interventions: Drug: anetumab ravtansine

INTERVENTIONS:
Drug: anetumab ravtansine — Patients will receive anetumab ravtansine IV infusion at a dose of 6.5 mg/kg (recommended Phase II dose) on Day 1 of a 21-day cycle

SUMMARY:
The primary objective of this study is to:

-Test the activity/response rate per RECIST 1.1 criteria of anetumab ravtansine in patients with advanced pancreatic cancer who stain for mesothelin expression

The secondary objectives of this study are to:

* Time to Progression (TTP) defined as time from study treatment to RECIST 1.1 progression, or death (others going off study will be censored)
* Toxicity in pancreatic cancer patients (at 6.5 mg/kg dose)

DETAILED DESCRIPTION:
This is a non-randomized, open-label, multicenter, Phase II study to evaluate the efficacy and safety of intravenous anetumab ravtansine (BAY 94-9343), an anti-mesothelin antibody drug conjugate, in pretreated mesothelin-expressing advanced pancreatic cancer.

At the time of the start of study treatment, the patients will have pretreated advanced pancreatic cancer that also overexpresses mesothelin as determined by immunohistochemistry (IHC).

A maximum of 30 patients will be enrolled in a minimax, Simon 2-stage design with a single early stopping rule for lack of efficacy. The target population is those patients with pancreatic cancer who have failed an earlier treatment. All patients will be treated with an anti-mesothelin immuno-conjugate, in this single arm, non-randomized trial and all patients treated with at least one dose of Anetumab will be included. The endpoint is any response using the RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for prescreening

* Must have had at least one and not more than two prior chemotherapy regimens for advanced disease (neoadjuvant or adjuvant chemotherapy would not be counted as a line of therapy). If prior radiation, measurable lesion outside radiation portal.
* Written informed consent for prescreening.
* Unresectable locally advanced or metastatic pancreatic cancer, confirmed by histology
* Availability of archival or fresh tissue for testing of mesothelin expression level.

Note: Archival tissue is preferred and fresh biopsy should only be obtained if no archival tissue is available and if in the investigator's judgement, there is no additional risk for the patient's safety. Patients with a sarcomatoid histology are not expected to have mesothelin overexpression and should not enter prescreening.

* Age ≥ 18 years.
* Life expectancy of at least 3 months.
* No prior treatment with anetumab ravtansine (or any other mesothelin-based therapy)

Eligibility criteria for full study

* Written informed consent for full study.
* Histological documentation of overexpressing mesothelin at the moderate (2+) or stronger (3+) level in at least 30% of tumor cells as determined by IHC.
* Unresectable locally advanced or metastatic pancreatic cancer
* At least one but not more than two prior chemotherapy regimens with progression or documented intolerance (neoadjuvant or adjuvant chemotherapy would not be counted as a line of therapy).
* Patients must have at least 1 measurable lesion according to RECIST v 1.1
* ECOG PS of 0 or 1
* Life expectancy of at least 3 months.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements conducted within 7 days before starting study treatment:
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN). Documented Gilbert syndrome is allowed if total bilirubin is mildly elevated (< 6 mg/dL).
* ALT and AST ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement of their cancer).
* ALP limit ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement of their cancer).
* Extent of baseline tumor burden will not interfere with causal assessment of treatment-emergent hepatotoxicity, at the investigator's discretion.
* Amylase and lipase ≤ 1.5 x ULN.
* Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2 according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula (see Appendix 16.6).
* Adequate coagulation, as assessed by the following laboratory test results:
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN (CTCAE Grade ≤ 1).
* Partial thromboplastin time (PTT) or activated PTT (aPTT) ≤ 1.5 x ULN (CTCAE Grade ≤ 1).

Note: Patients on stable dose of anti-coagulation therapy will be allowed to participate if they have no sign of bleeding or clotting and INR / PT and PTT / aPTT test results are compatible with the acceptable benefit-risk ratio at the investigator's discretion

* Platelet count ≥ 75,000/mm3 , without platelet transfusion within 3 weeks before the start of study treatment.
* Hemoglobin (Hb) ≥ 8 g/dL, without blood transfusion or erythropoietin within 6 weeks before the start of study treatment.

Note: Patients on stable dose of anti-coagulation therapy will be allowed to participate if they have no sign of bleeding or clotting and INR / PT and PTT / aPTT test results are compatible with the acceptable benefit-risk ratio at the investigator's discretion (see Section 8.1).

* Absolute neutrophil count (ANC) ≥ 1000/mm3
* Left ventricular ejection fraction (LVEF) ≥ 50% or the lower limit of normal (LLN) according to local institution ranges of normality

Exclusion Criteria:

* Previous assignment to treatment during this study. Patients permanently withdrawn from study participation will not be allowed to re-enter the study.
* Previous (within 5 drug half-lives - if drug half-life in subjects is known - or 28 days, whichever is shorter, before the start of study treatment) or concomitant participation in another clinical study with investigational medicinal product(s) (IMP[s]).
* Patients with corneal epitheliopathy or any eye disorder that may predispose the patients to this condition at the discretion of the investigator.
* Previous or concurrent cancer that is distinct in primary site or histology within 5 years. Exceptions: curatively treated
* Cervical cancer in situ.
* Non-melanoma skin cancer.
* Superficial bladder tumors (Non-invasive tumor [Ta], Carcinoma in situ [Tis] and Tumor invades lamina propria [T1]).
* Major surgery, open biopsy or significant traumatic injury within 28 days before the start of study treatment.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a serum pregnancy test performed a maximum of 7 days before the start of study treatment, and a negative result must be documented before the start of study treatment.
* Pre-existing cardiac conditions as outlined below:
* Congestive heart failure ≥ New York Heart Association (NYHA) class 2.
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months). Myocardial infarction less than 6 months before the start of study treatment.
* Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Clinically significant uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or venous pulmonary embolism within 6 months before the start of study treatment; venous thrombotic events such as deep vein thrombosis within 3 months before the start of study treatment.
* Ongoing or active infection (bacterial, fungal, or viral) of NCI-CTCAE version 4.03 Grade > 2.
* Known history of human immunodeficiency virus (HIV) infection.
* Known history of chronic hepatitis B or C.
* Patients with seizure disorder requiring medication.
* Symptomatic brain metastases or meningeal tumors or other uncontrolled metastases in the central nervous system (CNS) unless the patient
* Is > 6 months from definitive therapy,
* Has a negative imaging study within 4 weeks before study entry (ICF signature for full study) and
* Is clinically stable with respect to the tumor at the time of study entry.
* History of organ allograft, stem cells or bone marrow transplant.
* Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks before the start of study treatment.
* Non-healing wound, ulcer, or bone fracture.
* Renal failure requiring peritoneal dialysis or hemodialysis.
* Known hypersensitivity to anetumab ravtansine, study drug classes or excipients in the formulation.
* Any illness or medical conditions that are unstable or could jeopardize the safety of the patient and his/her compliance in the study.
* Unresolved toxicity higher than NCI-CTCAE version 4.03 Grade 1 attributed to any prior therapy/procedure excluding anemia or neuropathy Grade 2 and alopecia of any Grade.
* Any prohibited prior or concomitant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Stein, MD, Principal Investigator — Yale Cancer Center, Yale University
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 18
Completed | 14
Not Completed | 4
Not completed — No follow-up assessment | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 18
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 2
  60-69 years | 6
  70-79 years | 7
  80-89 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Response Rate as Measured Per RECIST 1.1 Criteria
Description: Primary efficacy will be assessed based on radiological tumor evaluation by contrast-enhanced computed tomography (CT) or contrast-enhanced magnetic resonance imaging (MRI) of chest/abdomen/pelvis. Contrast enhanced RECIST 1.1 scan will be done at Prescreening. Said pre-screen scan will be the baseline measure. RECIST 1.1 Scans will be done every 6 weeks for the first 6 months after the start of treatment, or more frequently if clinically indicated, every 9 weeks until the end of year 2 and every 12 weeks thereafter until disease progression or end of study, whichever comes first.
Time Frame: From start of treatment until disease progression or death (up to 3 years).
Population: Of the 18 subjects originally enrolled, the analysis population includes the 14 subjects who completed the study. The original intention was to follow subjects for up to 3 years. However, all subjects died before the three year mark, so the study was concluded on Dec. 11.2019, after 2 years and 7 months.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 14
Participants
  progressive disease | 12
  stable disease | 2

2. Secondary Outcome: Time to Progression
Description: Time to Progression (TTP) defined as time from study treatment to RECIST progression, or death (others going off study will be censored).
Time Frame: From start of treatment until disease progression or death (up to 3 years).
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | All Subjects
Number analyzed (Participants) | 14
days | 63.5 [22 to 148]

3. Secondary Outcome: Drug Toxicity
Description: Toxicity of Anetumab ravtansine assessed with National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. See adverse events for details. Participants who experienced any adverse events are included here.
Time Frame: From start of treatment until disease progression or death (up to 3 years).
Population: Detailed results are included under adverse events. The original intention was to follow subjects for up to 3 years. However, all subjects died before the three year mark, so the study was concluded on Dec. 11.2019, after 2 years and 7 months.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 18
Participants
  Serious adverse events: Yes | 11
  Serious adverse events: No | 7
  Other adverse events: Yes | 18
  Other adverse events: No | 0

ADVERSE EVENTS:
Time Frame: Three years.
Description: The original intention was to follow subjects for up to 3 years. However, all subjects died before the three year mark, so the study was concluded on Dec. 11.2019, after 2 years and 7 months.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 18/18
Serious Adverse Events (participants affected / at risk) | 11/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=18)
Fever (General disorders) | 1 (1) — Fever
Cognitive Disturbance (Nervous system disorders) | 1 (1) — Cognitive Disturbance
Stroke (Nervous system disorders) | 1 (1) — Stroke
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — Acute Kidney Injury
Hypotension (Vascular disorders) | 1 (1) — Hypotension
Obstruction Gastric (Gastrointestinal disorders) | 1 (1) — Obstruction Gastric
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Abdominal Pain
Ascites (Gastrointestinal disorders) | 1 (1) — Ascites
Sepsis (Infections and infestations) | 1 (1) — Sepsis
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dyspnea
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hypoxia
Palmar Plantar Erythrodysesthes (Skin and subcutaneous tissue disorders) | 1 (1) — Palmar Plantar Erythrodysesthes
Blood and Lymphatic System Disorders-other (Blood and lymphatic system disorders) | 1 (1) — Febrile Neutropenia
Infections and Infestations-other (Infections and infestations) | 1 (1) — Elevated White Blood Count
Respiratory Failure (Pleural metastatic PD) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory Failure (Pleural metastatic PD)
Constipation (Gastrointestinal disorders) | 1 (1) — Constipation
General Disorders and administration-other specify Failure to Thrive (General disorders) | 1 (1) — Failure to thrive
General Disorders and administration-other specify Death NOS (General disorders) | 1 (1) — Death NOS
Infections and Infestations-Other, specify-Rhinovirus (Infections and infestations) | 1 (1) — Rhino virus
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=18)
Abdominal distension (Gastrointestinal disorders) | 1 (1) — Abdominal distention
Abdominal pain (Gastrointestinal disorders) | 12 (19) — Abdominal Pain
Activated partial thromboplastin time prolonged (Cardiac disorders) | 3 (4) — PTT Prolonged
Acute kidney injury (Renal and urinary disorders) | 2 (2) — Aacute kidney injury
Alanine aminotransferase increased (Investigations) | 3 (4) — Alanine Aminotransferase Elevated
Alkaline phosphatase increased (Investigations) | 6 (7) — Alkaline Phosphatase Increase
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Allergic Rhinitis
Anemia (Blood and lymphatic system disorders) | 8 (12) — Anemia
Anorexia (Metabolism and nutrition disorders) | 11 (14) — Anorexia
Anxiety (Psychiatric disorders) | 5 (6) — Anxiety
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Arthralgias
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) — Arthritis - knees / hands
Ascites (Gastrointestinal disorders) | 2 (2) — Ascites
Aspartate aminotransferase increased (Investigations) | 2 (2) — AST Increase
Atrial fibrillation (Cardiac disorders) | 3 (4) — Atrial fibrillation
Atrial flutter (Cardiac disorders) | 1 (1) — Atrial flutter
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) — Back pain
Basal Cell Carcinoma of Skin (Skin and subcutaneous tissue disorders) | 1 (1) — Basal Cell Carcinoma of Skin
Bladder Cancer (Renal and urinary disorders) | 1 (1) — Bladder Cancer
Blood bilirubin increased (Investigations) | 3 (6) — Elevated bilirubin
Blurred vision (Eye disorders) | 3 (4) — Blurred Vison
Cardiac troponin I increased (Investigations) | 1 (1) — cardiac troponin i increased
Cataract (Eye disorders) | 1 (1) — Cataracts
Chills (General disorders) | 3 (4) — Chills
Cholesterol high (Investigations) | 1 (1) — High Cholesterol
Constipation (Gastrointestinal disorders) | 11 (19) — Constipation
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dry Cough
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Cough
Creatinine increased (Investigations) | 1 (4) — Creatinine Increase
Decreased Platelet Count (Blood and lymphatic system disorders) | 1 (1) — Decreased Platelet Count
Dehydration (Metabolism and nutrition disorders) | 5 (8) — Dehydration
Depression (Psychiatric disorders) | 4 (5) — Depression
Diabetes (Metabolism and nutrition disorders) | 3 (3) — diabetes
Diarrhea (Gastrointestinal disorders) | 10 (16) — Diarrhea
Dizziness (Nervous system disorders) | 3 (3) — Dizziness
Dry eye (Eye disorders) | 7 (7) — Dry Eyes
Dry mouth (Gastrointestinal disorders) | 2 (2) — Dry Mouth
Dysgeusia (Nervous system disorders) | 1 (1) — Dysgeusia
Dyspepsia (Gastrointestinal disorders) | 3 (4) — Dyspepsia
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dyspnea
Edema limbs (General disorders) | 5 (7) — Edema limbs
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 2 (3) — Prolonged QTC
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) — Facial Erythema
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Colorblindness
Eye pain (Eye disorders) | 1 (1) — Right eye pain
Fall (Injury, poisoning and procedural complications) | 1 (1) — Fall
Fatigue (General disorders) | 14 — Fatigue
Fever (General disorders) | 2 (3) — fevers
Flatulence (Gastrointestinal disorders) | 1 (1) — Flatulence
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3) — GERD
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Partial gastric outlet obstruction
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Abdominal hernia
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — Mouth sores
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Generalized muscle weakness
GGT increased (Investigations) | 1 (1) — GGT increased
Glaucoma (Eye disorders) | 1 (1) — Glaucoma
GOUT (Metabolism and nutrition disorders) | 1 (1) — GOUT
Headache (Nervous system disorders) | 1 (2) — Headache
Hearing impaired (Ear and labyrinth disorders) | 1 (1) — Hearing impaired
Hematuria (Renal and urinary disorders) | 1 (1) — Hematuria
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hiccups
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hoarseness
Hypercholesterolemia (Investigations) | 1 (1) — Hypercholesterolemia
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — hyperglycemia
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — Hypokalemia
Hypertension (Vascular disorders) | 7 (17) — Hypertension
Hypertriglyceridemia (Blood and lymphatic system disorders) | 1 (1) — Hyperlipidemia
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4) — Hyperuricemia
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6) — Hypoalbuminemia
Hypocalcemia (Metabolism and nutrition disorders) | 3 (6) — Hypocalcemia
Hypokalemia (Metabolism and nutrition disorders) | 3 (8) — Hypokalemia
hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) — Hypomagnesemia
Hyponatremia (Metabolism and nutrition disorders) | 4 (5) — Hyponatremia
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) — Hypophosphatemia
Hypotension (Vascular disorders) | 1 (2) — Orthostatic Hypotension
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hypoxia
Increased LDH (Investigations) | 1 (1) — Increased LDH
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Oral Thrush
Inguinal hernia (Gastrointestinal disorders) | 1 (1) — inguinal hernia
INR increased (Investigations) | 4 (5) — Elevated INR
Insomnia (Psychiatric disorders) | 9 (12) — Insomnia
Investigations - Other, specify (Nervous system disorders) | 1 (1) — Tremors
Investigations- other, specify (Investigations) | 1 (1) — Elevated LDH
Irritability (General disorders) | 1 (1) — Irritability
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) — Left Ventricular Systolic Dysfunction
Lipase (Investigations) | 1 (1) — Lipase
Lymphocyte count decreased (Investigations) | 5 (9) — lymphocyte count decrease
Malabsorption (Gastrointestinal disorders) | 1 (1) — Malabsorption
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — Decreased appetite
Mucositis oral (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Mucositis
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) — myalgia
Nausea (Gastrointestinal disorders) | 9 (18) — Nausea
Neuropathy (Nervous system disorders) | 1 (1) — Neuropathy
Non-cardiac chest pain (General disorders) | 1 (1) — Non cardiac chest pain
Occasional Epigastric Pain (Gastrointestinal disorders) | 1 (1) — Occasional Epigastric Pain
Orthostatic Hypotension (Vascular disorders) | 1 (2) — Orthostatic Hypotension
Pain (General disorders) | 1 (1) — Pain (back/neck)
Paresthesia (Nervous system disorders) | 1 (1) — Bilateral Hands
Peripheral sensory neuropathy (Nervous system disorders) | 8 (12) — Peripheral Sensory Neuropathy
Platelet count decreased (Investigations) | 4 (7) — platelet count decrease
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) — Pleural effusion
Proteinuria (Renal and urinary disorders) | 5 (8) — Proteinuria
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Pruritis
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) — Mood Swings
Rash (Skin and subcutaneous tissue disorders) | 1 (2) — Rash
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (3) — Kidney stone
Serum amylase increased (Investigations) | 1 (1) — Serum Amylase Increased
Sick sinus syndrome (Cardiac disorders) | 1 (1) — Sick Sinus Syndrome
Sinus tachycardia (Gastrointestinal disorders) | 2 (4) — Sinus Tachycardia
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Sleep apnea
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) — small intestinal obstruction
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Sore Throat
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) — Thrombocytopenia
Upper respiratory infection (General disorders) | 1 (1) — Cold
URI/ Sinus Symptoms (Infections and infestations) | 1 (1) — URI/ Sinus Symptoms
Urinary frequency (Renal and urinary disorders) | 1 (1) — Urinary Frequency
Urinary retention (Renal and urinary disorders) | 1 (1) — urinary retention
Urinary tract infection (Infections and infestations) | 1 (1) — Urinary tract infection
Vomiting (Gastrointestinal disorders) | 9 (13) — Vomiting
Watering eyes (Eye disorders) | 1 (1) — Watering Eyes
Weight loss (Gastrointestinal disorders) | 4 (5) — Weight Loss
White blood cell decreased (Investigations) | 1 (1) — WBC Count Decrease

LIMITATIONS AND CAVEATS:
Premature termination may occur if risk-benefit ratio is unacceptable due to: safety findings, results of parallel clinical studies and results of parallel animal studies AND if the study does not suggest a completion within a reasonable time frame.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT03023722/Prot_SAP_000.pdf